CLINICAL TRIAL: NCT01262573
Title: Barbed Suture vs Smooth Suture for Vaginal Cuff Closure, a Randomized Trial
Brief Title: Barbed Suture vs Smooth Suture for Vaginal Cuff Closure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jon I. Einarsson, Chief, Division of Minimally Invasive Gynecology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010P001586
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Closure of Vaginal Cuff at Laparoscopic Hysterectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Barbed (Experimental): Vaginal cuff closure with barbed suture
  Interventions: Procedure: Closure of vaginal cuff
- Smooth (Active Comparator): Vaginal cuff closure with smooth suture
  Interventions: Procedure: Closure of vaginal cuff

INTERVENTIONS:
Procedure: Closure of vaginal cuff — Closure of the vaginal cuff

SUMMARY:
This study compares outcomes among patients having a total laparoscopic hysterectomy. This involves removing the uterus and cervix using a laparoscopic or keyhole technique. The top of the vagina is routinely sutured closed after this procedure and this study is comparing two different suture materials for this purpose. One suture material is a barbed suture that has the advantage of maintaining good tension and closure on the wound. The other is a standard smooth suture that is commonly used for this procedure. The investigators are comparing the time it takes to close the vaginal cuff, as well as bleeding after surgery and the healing of the top of the vagina.

DETAILED DESCRIPTION:
Barbed suture has been used to close the vaginal vault for almost 3 years now, and a few preliminary studies report positive outcomes. Unfortunately, the retrospective nature of these studies may present outcomes in an overly positive light, since some of the patients may not be able to remember all the potential complications or problems they may have had in the immediate postoperative period (recall bias). The current standard of care for vaginal cuff closure appears to be to use Vicryl suture although practices vary widely.

The specific aim of this study is to evaluate whether the use of barbed suture facilitates the laparoscopic closure of the vaginal cuff during a total laparoscopic hysterectomy.

The inclusion criteria for our study include all patients who are planned for a total laparoscopic hysterectomy due to benign conditions such as symptomatic uterine fibroids, abnormal uterine bleeding, endometriosis and pelvic pain.

The laparoscopic hysterectomy will proceed as per routine. For vaginal cuff closure with barbed suture we will use a 0 polydioxanone (PDO) bidirectional barbed suture on a 36 mm half-circle taper point needle. For cuff closure with Vicryl, we plan to use 2/0 Vicryl with the vaginal cuff closure proceeding in a similar fashion as with the barbed suture. Regardless of suture material used it is important to obtain a full thickness bite with a 1 cm margin on the vagina mucosa on each bite.

Patients will be stratified to either closure by the attending or the resident or fellow under the supervision of the attending. The resident or fellow will have 15 minutes to complete the vaginal cuff closure. If they are not able to complete it within that time frame, the attending will take over and complete the vaginal cuff closure. This is to avoid adding excess operating time to the procedure due to having a trainee performing a portion of the procedure. Patients will also be asked to complete a short survey regarding dyspareunia as well as a standardized sexual function questionnaire (FSFI) prior to surgery and 3 months after surgery to evaluate if the use of barbed suture affects this in any way. Further we will also inquire about male dyspareunia before and after surgery for the same reason.

Patients will be examined at a postoperative visit 3 weeks after surgery and vaginal cuff granulation and any evidence of vaginal cuff infection or separation will be carefully examined and documented. Patients will be called 3 months after surgery to inquire about any dyspareunia, male dyspareunia, vaginal bleeding or readmissions to the hospital. We are interested in evaluating dyspareunia, since a concern has been raised that the use of barbed suture at the vaginal apex may result in dyspareunia and partner dyspareunia. Although we have not found this to be the case in our clinical experience we would like to evaluate this point, especially since the use of barbed suture for closing the vaginal cuff has become a common practice nationwide. Patients will be dismissed from the trial after the 3 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a total laparoscopic hysterectomy for benign conditions

Exclusion Criteria:

* Malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Barbed | Smooth
Started | 32 | 32
Completed | 32 | 31
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Barbed | Smooth | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (5.6) | 43.2 (8.1) | 44.7 (0.71)
Gender [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 19 | 19 | 38
  Black | 8 | 8 | 16
  Hispanic | 2 | 2 | 4
  Asian | 2 | 1 | 3
  Other | 0 | 1 | 1
  Unknown | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 63
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.1 (5.9) | 26.9 (8.6) | 28.0 (4.2)
Parity [Mean (Standard Deviation); unit: Births] | 1.7 (1.3) | 1.7 (1.0) | 1.7 (0)
Smoking Status - Smoker [Number; unit: participants] | 2 | 7 | 9
Marital Status - Married [Number; unit: participants] | 11 | 12 | 23
Hospital [Number; unit: participants]
  Brigham and Women's Hospital | 11 | 11 | 22
  Faulkner Hospital | 7 | 7 | 14
  Army Hospital | 14 | 13 | 27
Cuff closure performed by the Attending Surgeon or the Fellow/Resident [Number; unit: participants]
  Attending | 16 | 15 | 31
  Fellow/Resident | 16 | 16 | 32
Medical History [Number; unit: participants]
  Fibroids | 21 | 20 | 41
  Pelvic Pain | 23 | 24 | 47
  Infertility | 3 | 2 | 5
  Prolapse | 0 | 0 | 0
  Abnormal Uterine Bleeding | 27 | 24 | 51
  Prior Laparoscopy | 15 | 12 | 27
  Prior Laparotomy | 12 | 19 | 31
Sexual Function [Number; unit: participants]
  Any female dyspareunia reported | 12 | 13 | 25
  Any male dyspareunia reported | 0 | 0 | 0
  Ongoing problem | 5 | 0 | 5
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Vaginal Cuff Closure Time
Description: Average time (measured in minutes)
Time Frame: During the surgical procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Barbed | Smooth
Number analyzed (Participants) | 32 | 31
minutes | 10.4 (5.2) | 9.6 (4.8)

2. Secondary Outcome: Dyspareunia
Description: Assessed preoperatively and up to 3 months postop
Time Frame: Postoperative
Measure: Number; unit: participants
Arm/Group | Barbed | Smooth
Number analyzed (Participants) | 32 | 31
participants
  Any female dyspareunia reported | 2 | 1
  Any male dyspareunia reported | 1 | 0
  Ongoing problem | 0 | 1
  Other | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 3 months after surgery
Arm/Group | Barbed | Smooth
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes